CLINICAL TRIAL: NCT01701531
Title: An Open-Label, Pilot Study of a Red Blood Cell Precursor Formulation to Determine Increased Production in Subjects With Mild to Moderate Anemia
Brief Title: Red Blood Cell Precursor Formulation to Determine Increased Production
Acronym: RBCPF
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding not received
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBC100312
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

ARMS (1):
- RBCPF (Experimental): Treatment intervention arm
  Interventions: Drug: RBCPF

INTERVENTIONS:
Drug: RBCPF
  Other Names: Red blood cell precursor formulation

SUMMARY:
The objective of this study is to measure the change in hemoglobin levels after the administration of an amino acid based, RBC precursor formulation.

DETAILED DESCRIPTION:
Medical foods are a distinct FDA regulatory category different from single molecule chemical pharmaceuticals, and from dietary supplements. The FDA has regulated amino acid preparations as drugs since the 1940s as they can elicit pharmacologic effects similar to conventional single molecule pharmaceuticals. The best known amino acid preparations are used to treat conditions such as maple syrup disease and phenylketonuria (PKU). An official definition and categorization of medical foods was made in 1988 as part of the Orphan Drug Act. Medical foods are regulated similarly to drugs except they do not require pre-approval because all ingredients are found on the FDA's generally recognized as safe (GRAS) (Sections 201(s) and 409 of the Federal Food, Drug, and Cosmetic Act) list and claims are confined to the nutritional management of a specific disease. Medical food claims must be supported by recognized scientific data as determined by medical evaluation. A GRAS substance is distinguished from a food additive on the basis of the common knowledge about the safety of the substance for its intended use. The standard for an ingredient to achieve GRAS status requires not only technical demonstration of non-toxicity and safety, but also general recognition of safety through widespread usage and agreement of that safety by experts in the field. Many ingredients have been determined by the FDA to be GRAS, and are listed as such by regulation, in Volume 21 Code of Federal Regulations (CFR) Sections 182, 184, and 186.

ELIGIBILITY:
Inclusion Criteria:

1. M/F patients 18 to 75 years old, non-pregnant/lactating
2. Male patients with < Hemoglobin of 12.5
3. Female Patients with < Hemoglobin of 11
4. Diagnosis of mild to moderate anemia by study physician

Exclusion Criteria:

1. Pregnant or unwilling to use adequate birth control for the duration of the study.
2. Unwilling or unable to sign informed consent.
3. Myocardial infarction within the last 6 months.
4. Patients currently taking an erythropoietin medication and unable to discontinue for the duration of the study.
5. GI bleed in the last 6 months.
6. Inflammatory bowel disease.
7. Chronic liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin level 2 hours after administration of the first dose. | Baseline, 2 hours and 7 days
  Subjects will have blood drawn at baseline and 2 hours after the administration of the treatment intervention. Then again, after 7 days.

SECONDARY OUTCOMES:
CBC w/ differential | Baseline, 2 hours and 7 days
Erythropoietin level | Baseline, 2 hours and 7 days
Reticulocytes | Baseline, 2 hours and 7 days
Iron levels | Baseline, 2 hours and 7 days
Ferritin | Baseline, 2 hours and 7 days
IGG | Baseline, 2 hours and 7 days
B12 | Baseline, 2 hours and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence May, MD, Principal Investigator — Lawrence May MD, Inc
Locations (1):
- Lawrence May, MD, Inc., Tarzana, California, United States